CLINICAL TRIAL: NCT02675439
Title: A Phase I, Open Label, Multicenter Study of the Safety and Efficacy of MIW815 (ADU-S100) Administered by Intratumoral Injection to Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Brief Title: Safety and Efficacy of MIW815 (ADU-S100) +/- Ipilimumab in Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No substantial anti-tumor activity was observed.
Sponsor: Chinook Therapeutics, Inc. (formerly Aduro) (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Chinook Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-07
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Advanced/Metastatic Solid Tumors or Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — ADU-S100; Ipilimumab

ARMS (2):
- Dose escalation monotherapy (Experimental): ADU-S100 administered intratumorally on Days 1, 8 and 15 of each 28-day cycle until unacceptable toxicity, progressive disease and/or treatment is discontinued; starting dose 50 micrograms
  Interventions: Drug: ADU-S100
- Dose escalation combination (Experimental): ADU-S100 administered intratumorally on Days 1 and 8 of each 21-day cycle (starting dose 200 micrograms) and ipilimumab, i.v., (3 mg/kg) on day 1 of each 21-day cycle for the first 4 cycles. Dosing is continued until unacceptable toxicity, progressive disease and/or treatment is discontinued
  Interventions: Drug: ADU-S100; Biological: ipilimumab

INTERVENTIONS:
Drug: ADU-S100
  Other Names: MIW815
Biological: ipilimumab
  Arms: Dose escalation combination

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics and antitumor activity of MIW815 (ADU-S100) administered via intratumoral injection as a single agent and in combination with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* ECOG ≤ 1
* Willing to undergo tumor biopsies from injected and distal lesions
* Must have two biopsy accessible lesions:

  * * one lesion must be ≥10 mm and <100 mm in longest diameter, accessible for repeated intratumoral (IT) injection and accessible for baseline and on-treatment biopsies.

    * a second (distal) lesion must be accessible for baseline and on-treatment biopsy and must be distinct from the injected lesion.
    * tumors encasing major vascular structures (i.e., carotid artery or tumors close to other vital organs), are not considered appropriate

Exclusion Criteria:

* Patients who require local palliative measures such as XRT or surgery
* Symptomatic or untreated leptomeningeal disease.
* Presence of symptomatic central nervous system (CNS) metastases
* Impaired cardiac function or clinically significant cardiac disease
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy.
* Active infection requiring systemic antibiotic therapy.
* Known history of Human Immunodeficiency Virus (HIV) infection.
* Active Epstein-Barr virus (EBV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Malignant disease, other than that being treated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Safety: Number of patients reporting treatment-related adverse events that qualify as dose-limiting toxicities | 6 months from study start
  Number of patients reporting treatment-related adverse events that qualify as dose-limiting toxicities
Recommended dose | 6 months from study start
  Using maximum tolerated dose to identify the recommended dose for future studies

SECONDARY OUTCOMES:
Pharmacokinetics measured through plasma concentrations | 6 months from study start
  measured through plasma concentrations
measurement of CD8-TIL counts | 6 months from study start
RNA expression analysis of IFN gamma and immunomodulatory genes | 6 months from study start

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center-Herbert Irving Pavilion, New York, New York
  - University of Texas/MD Anderson Cancer Center MD Anderson PSC, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Gogoi H, Mansouri S, Jin L. The Age of Cyclic Dinucleotide Vaccine Adjuvants. Vaccines (Basel). 2020 Aug 13;8(3):453. doi: 10.3390/vaccines8030453. PMID 32823563